CLINICAL TRIAL: NCT02694250
Title: Evaluation of Cervical Fusion With DTRAX® Cervical Cage With DTRAX Bone Screw in Patients With Cervical Radiculopathy
Brief Title: Evaluation of Cervical Fusion With DTRAX® Cervical Cage With DTRAX Bone Screw
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not started due to lack of resources
Sponsor: Providence Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTRAXCCB-001
Record Dates: First submitted 2016-02-15; First posted 2016-02-29 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cervical Radiculopathy
Keywords: cervical; fusion; radiculopathy; DTRAX
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DTRAX Cervical Cervical Cage with DTRAX Bone Screw (Other)
  Interventions: Device: DTRAX® Cervical Cage with DTRAX Bone Screw

INTERVENTIONS:
Device: DTRAX® Cervical Cage with DTRAX Bone Screw — DTRAX Cervical Cage is an intervertebral fusion device that provides mechanical support to the spine. DTRAX Cervical Cage is intended to be used in cervical spine fusion surgery. DTRAX Bone Screw is indicated for use in arthrodesis and provides supplemental fixation. .

SUMMARY:
This study is being conducted to assess the radiographic (x-rays and CT scans) and clinical outcomes for the use of DTRAX Cervical Cage with DTRAX Bone Screw for the treatment of degenerative disc disease at one disc level with accompanying radicular symptoms in the cervical (neck) spine.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with one level cervical spondylosis with radiculopathy in C3-C7, defined as follows:

   a. Radiographically (at least one): i. degenerated disc on MRI and/or CT; ii. decreased disc height on MRI and/or CT; and/or iii. foraminal stenosis, as demonstrated by MRI and/or CT. b. Clinically: radicular symptoms (at least one): i. arm/shoulder pain; ii. decreased reflexes; iii. decreased strength; and/or iv. decreased sensation.
2. Subject has dynamic stenosis relieved by traction and made worse by a Spurlings maneuver.
3. Subject is 35-80 years of age, inclusive.
4. Subject is unresponsive to 6 weeks conservative, nonoperative treatment, or clinically indicated sooner due to the presence of progressive symptoms or signs of nerve root in spite of combined nonoperative management.
5. Preoperative Neck Disability Index (NDI) score of > 30.
6. Preoperative Neck pain or Arm pain score of > 6 on Neck and Arm VAS Pain Scales.
7. Subject is a male or non-pregnant, non-lactating female.
8. Subject must have the ability to understand and voluntarily provide written, informed consent.
9. Subject is able to meet the proposed follow-up schedule.
10. Subject is able to follow the postoperative management program.

Exclusion Criteria:

1. Any previous cervical spinal surgery.
2. Subject has known osteoporosis, osteomalacia, spinal metastases, or metabolic bone disease OR subject has sustained a vertebral compression or nontraumatic hip or wrist fracture.
3. Subject has overt or active spinal and/or systemic infection.
4. Subject has cervical spondylolisthesis > 3.5mm or rotator subluxation.
5. Subject has cervical myelopathy.
6. Subject has a chronic pain syndrome.
7. Subject has radicular findings with major motor impairment.
8. Subject has a condition that requires postoperative medications that interfere with fusion or the stability of the implant, such as steroids (ie. corticosteroids, methotrexate, immunosuppressives).
9. Subject is mentally incompetent.
10. Subject is a prisoner.
11. Subject is pregnant.
12. Subject abuses alcohol or drugs.
13. Subject has a cervical spinal condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level.
14. Subject has insulin dependent diabetes.
15. Subject has chronic or acute renal failure or prior history of renal disease.
16. Subject has documented allergy or intolerance to stainless steel, titanium, or a titanium alloy.
17. Subject has or is planning to receive drugs which may interfere with bone metabolism within two weeks prior to or six months following the date of surgery.
18. Subject has history of an endocrine or metabolic disorder known to affect osteogenesis.
19. Subject has had treatment with an investigational therapy within 28 days prior to surgery or such treatment is planned during the 16 weeks following implantation of DTRAX Cervical Cage with DTRAX Bone Screw.
20. Subject is involved in or planning spinal litigation or Workmen's Compensation claim.
21. Subject is morbidly obese, defined as body mass index (BMI) > 40.
22. Subject has a medical condition or extenuating circumstance that, in the Investigator's opinion, would prevent the subject from complying with postoperative follow-up visits.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Assess the radiographic outcome data on fusion status, device retention, and maintenance of segmental lordosis at the index level utilizing DTRAX Cervical Cage with DTRAX Bone Screw used in the treatment of cervical radiculopathy | Baseline throughout 24 months post-operatively

SECONDARY OUTCOMES:
Assess the clinical outcome data based Neck Disability Index (NDI) | Baseline throughout 24 months post-operatively
Assess the clinical outcome data based SF-12 v2 Health Survey | Baseline throughout 24 months post-operatively
Assess the clinical outcome data based the Visual Analogue Scale (Neck and Arm VAS) | Baseline throughout 24 months post-operatively
Safety information will be evaluated by collecting the type, frequency, severity, and device and procedure-relatedness of adverse events | Baseline throughout 24 months post-operatively

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Neurospine Institute Medical Group, San Francisco, California
  - Daytona Orthopaedic and Spinal Research Group, Daytona Beach, Florida
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Louisiana State University Health Sciences Center - New Orleans (LSUHSC - NO), New Orleans, Louisiana
  - Upstate Orthopedics, East Syracuse, New York
  - Southern New York NeuroSurgical Group, P.C., Johnson City, New York
  - Cary Orthopaedic Spine Specialists, Cary, North Carolina

IPD SHARING:
Plan to Share IPD: No